CLINICAL TRIAL: NCT04246918
Title: Effect of Branched Chain Amino Acids Supplementation on Muscle Mass, Muscle Quality and Molecular Markers of Muscle Regeneration in Patients With Chronic Liver Disease - A Randomized Controlled Trial.
Brief Title: Effect of BCAA Supplementation on Muscle Mass, Muscle Quality and Molecular Markers of Muscle Regeneration in CLD Patients
Acronym: BCAA-CLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-BCAA-02
Record Dates: First submitted 2020-01-20; First posted 2020-01-29 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2022-03

CONDITIONS: Chronic Liver Disease
Keywords: Chronic Liver Disease; Sarcopenia; Myostatin; Health related quality of life; muscle histology
MeSH Terms: conditions — Sarcopenia | interventions — Amino Acids, Branched-Chain

STUDY DESIGN:
Intervention Model Description: Open Label
Masking Description: As it is a nutritional intervention study masking either the participant or the investigator is not possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Treatment Group (Placebo Comparator): The patients would receive customized diet charts providing 30-35Kcal/ideal body wt/day and 1.5 gm protein/ideal body wt/day) describing the food items along with the quantity and approximate household measurements. Diet would be so planned for each patient keeping in mind the individual food habits and choices. This group would not receive any supplement other than the prescribed diet. Whey protein will be included in this group.
  Interventions: Dietary Supplement: Whey Protein concentrate powder
- Intervention Arm (Active Comparator): The patients would receive customized diet charts providing 30-35Kcal/ideal body wt/day and 1.5 gm protein/ideal body wt/day) describing the food items along with the quantity and approximate household measurements. Diet would be so planned for each patient keeping in mind the individual food habits and choices. In addition to the normal diet this group would receive 16gm of branched chain amino acid (BCAA) supplement (Commercial oral BCAA granules) daily in 4 divided doses, keeping the protein levels within the same range of 1.5 gm/Kg/day.
  Interventions: Dietary Supplement: Branched Chain Amino Acid

INTERVENTIONS:
Dietary Supplement: Branched Chain Amino Acid — Branched chain amino acid is a group of three amino acids known for there role in muscle growth.
  Arms: Intervention Arm
Dietary Supplement: Whey Protein concentrate powder — Whey protein will be given to the standard treatment arm including in the same amount of 1.5gm/kg/IBW.
  Arms: Standard Treatment Group

SUMMARY:
Loss of muscle mass (sarcopenia) is a major complication in a patient with cirrhosis, impacting the disease outcome, quality of life and survival. Cirrhotics lose muscle mass (MM) while waiting for liver transplant (LT) and even after LT, impacting the outcome of LT. Moreover, LT is elusive for majority of patients in India. The pathophysiology of muscle loss is complicated, multifactorial, interlinked and primarily nutrition driven, which gives clues for targeted therapeutic modalities other than feeding alone. Experimental studies have instilled faith in BCAA in successfully counteracting the pathogenesis of muscle loss. But there is lack of convincing data from clinical studies with direct evidence on muscle growth per se.

DETAILED DESCRIPTION:
Reduction in muscle mass (sarcopenia) is well documented in patients with chronic liver disease (CLD)leading to increased morbidity, mortality and poor quality of life. An equilibrium is maintained between the synthesis and degradation of muscles to maintain the muscle mass. However, an imbalance between the synthesis and degradation leads to loss of muscle mass. Various factors like alteration in dietary intake, hyper-metabolism, changes in amino acid profile, decreased physical activity, endotoxemia, hyperammonemia, increased myostatin levels have been postulated in the pathogenesis of muscle loss in liver disease. Reduced dietary intake, altered amino acid profile, decreased physical activity down regulate the anabolic pathway while the others increase the catabolic pathway. Increased level of myostatin inhibits the mTOR signaling and increases catabolism. Various therapeutic strategies such as increased calorie and protein intake, branched chain amino acid (BCAA) supplementation, late evening snack (LES), increased physical activity are the well accepted therapies. Hormone therapy (testosterone/growth hormone) also has been tried to improve muscle mass and function, reduce muscle catabolism in patients with CLD, however these newer treatment modalities i.e. hormone replacement, immune-nutrition and anti-myostatin antibodies are not free from adverse side-effects. Branched chain amino acids, a group of three essential amino acids (leucine, isoleucine, valine) have been tried since years in the setting of chronic liver disease patients for the treatment of hepatic encephalopathy and improvement in nutritional status. However, the studies assessing the impact of nutrition and BCAA in CLD have not assessed the direct impact on the muscle per se. The nutritional status has been assessed using different subjective methods like mid arm muscle circumference, triceps skin fold, nitrogen balance. Nutritional management is the cornerstone of the overall management of patients with cirrhosis, wherein BCAA constitutes an important therapeutic modality in the realm of nutrition in liver disease.

In the present study all the eligible cirrhotic patients will be randomized to a control group (receiving the nutritional therapy as per the standard nutritional practices and guidelines) or the intervention group (receiving BCAA supplementation over and above the standard nutrition therapy as per the standard nutritional practices and guidelines). Branched chain amino acids (BCAA) have the potential to up-regulate the anabolic pathway of muscle synthesis leading to improvement in muscle mass. Muscle mass as assessed by DEXA, along with changes in muscle histology, markers of the pathways that regulate muscle growth, functional capacity, and quality of life will be assessed after 3 months of BCAA intervention.

ELIGIBILITY:
Inclusion Criteria:

* Patients with decompensated cirrhosis (CTP 7-9)
* Adult patients Age 18-60 years
* Patients with corrected BMI in the range <22.9
* Those who give consent for muscle biopsy
* INR <1.5 or 1.5-2.5 after correction with Vitamin K
* Platelets > 80000
* All etiologies

Exclusion Criteria:

* Presence of overt hepatic encephalopathy
* Patients with co-morbidities e.g. acquired immunodeficiency syndrome, HCC, Other cancer, Diabetes Mellitus, chronic kidney disease, congestive heart disease , chronic respiratory disease
* Patients with alcohol intake in past 3 months
* Patients with TIPS
* Patients on steroids
* INR >2.5
* Refusal to participate in the trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Improvement in the muscle mass | 3 months
  Muscle mass change as assessed by DEXA scan will be done.

SECONDARY OUTCOMES:
Changes in the muscle fibre type composition | 3 months
  Muscle fibre type will be assessed in muscle biopsy sample
Changes in cross sectional area of muscle | 3 months
  Muscle fibre cross sectional area will be assessed in muscle biopsy sample
Assessment of necrosis in muscle fibre | 3 Months
  Muscle fibre necrosis will be assessed in muscle biopsy sample
Assessment of intramuscular fat deposition | 3 months
  Change in intramuscular fat deposition will be assessed in muscle biopsy sample.
Assessment of myoD | 3 month
  Change in myoD will be assessed as marker of muscle regeneration in muscle biopsy sample
Assessment of myogenin | 3 months
  Change in myogenin will be assessed as marker of muscle regeneration in muscle biopsy sample
Assessment of PCNA | 3 months
  Change in PCNA as marker of satellite function will be assessed in muscle biopsy sample
Assessment of proteosome C3, C5, C9 | 3 months
  Change in these proteosome will be assessed in muscle biopsy sample
Assessment of ubiquitin ligase E3 | 3 months
  Change in Ubiquitin ligase E3 will be assessed in muscle biopsy sample.
Assessment of myostatin level | 3 months
  Change in myostatin level will be assessed in blood sample using commercially available kit.
Assessment of ammonia level | 3 months
  Change in ammonia level will be assessed in blood sample using commercially available kit
Assessment of Insulin resistance | 3 Month
  Insulin resistance will be calculated using homeostasis model for insulin resistance.
Assessment of IGF 1 | 3 Month
  IGF1 will be assessed using commercially available kit.
Assessment of Nutritional Status | 3 Month
  Change Nutritional status will be assessed using bioelectrical impedance analysis
Assessment of Nitrogen balance | 3 Month
  Change in nitrogen balance will be assessed using formula : Nitrogen Balance = Protein intake (gm) / 6.25 - (UUN + 4 gm)
Assessment of functional capacity | 3 Months
  The Functional capacity of the patients would be assessed by Hand Grip Strength using the Handgrip Dynamometer .
Assessment of Clinical parameter- CTP | 3 Months
  Clinical improvement will be assessed in terms of change in CTP score.
Assessment of Clinical parameter-MELD | 3 Months
  Clinical improvement will be assessed in terms of change in MELD score.
Assessment of Health Related Quality of Life | 3 Months
  The Health Related Quality of Life (HRQoL) of the patients would be assessed using the Chronic liver disease questionnaire(CLDQ)

CONTACTS AND LOCATIONS:
Overall Officials: Puja Bhatia, MSc, Principal Investigator — Institute of Liver and Biliary Sciences; Jaya Benjamin, PhD, Study Director — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India